CLINICAL TRIAL: NCT04494828
Title: Impact of Prophylactic Use of Dexmedetomidine on Postoperative Delirium in Patients After Intracranial Operation for Brain Tumor: a Pilot Randomized Controlled Trial
Brief Title: Impact Dexmedetomidine on Postoperative Delirium in Patients After Intracranial Operation for Brain Tumor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2019-091-02A
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Central Nervous System Diseases
Keywords: delirium; postoperative; dexmedetomidine; intracranial operation; prevention
MeSH Terms: conditions — Central Nervous System Diseases; Delirium | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Continuously intravenous infusion of dexmedetomidine hydrochloride at a rate of 0.1 μg/ kg/hour (0.025 ml/kg/hour) started immediately after enrollment until 08:00 AM on the postoperative day one.
  Interventions: Drug: Dexmedetomidine
- Normal saline group (Placebo Comparator): Continuously intravenous infusion of normal saline at a rate of 0.025 ml/kg/hour started immediately after enrollment until 08:00 AM on the postoperative day one.
  Interventions: Drug: Normal saline group

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine hydrochloride (200 μg/2 ml) is diluted with normal saline to 50 ml and is continuously intravenous infused at a rate of 0.025 ml/kg/hour (dexmedetomidine 0.1 μg/kg/hour). The intravenous infusion begins immediately after enrollment until 08:00 AM on the postoperative day one.
  Other Names: Dexmedetomidine hydrochloride
  Arms: Dexmedetomidine group
Drug: Normal saline group — Normal saline is also diluted with normal saline to 50 ml and is continuously intravenous infused at a rate of 0.025 ml/kg/hour, which is the same with the dexmedetomidine group. The intravenous infusion begins immediately after enrollment until 08:00 AM on the postoperative day one.
  Other Names: 0.9% Sodium Chloride
  Arms: Normal saline group

SUMMARY:
Postoperative delirium is one of the most common serious complications after major surgery and is associated with undesirable consequences. Prevention of postoperative delirium is recommended in the clinical guidelines and consensus statements. Dexmedetomidine, a highly selective α2-adrenergic receptor agonist, has been investigated as a pharmacological intervention to prevent postoperative delirium. Several randomized controlled trials have shown that prophylactic use of low-dose dexmedetomidine may decrease the incidence of postoperative delirium in patients after cardiac and non-cardiac operations. However, neurosurgical patients are often excluded from previous studies due to potential consciousness and cognition impairment. The investigators design this pilot study aiming to clarify the feasibility and safety of use of low-dose dexmedetomidine for prevention of postoperative delirium in patients after intracranial operation for brain tumor.

DETAILED DESCRIPTION:
Postoperative delirium is one of the most common serious complications after major surgery and is associated with undesirable consequences. Prevention of postoperative delirium is recommended in the clinical guidelines and consensus statements. Dexmedetomidine, a highly selective α2-adrenergic receptor agonist, has been investigated as a pharmacological intervention to prevent postoperative delirium. Several randomized controlled trials have shown that prophylactic use of low-dose dexmedetomidine (0.1 ug/kg/hour without loading infusion) may decrease the incidence of postoperative delirium in patients after cardiac and non-cardiac operations. However, neurosurgical patients are often excluded from previous studies due to potential consciousness and cognition impairment. The investigators design this pilot randomized controlled trial aiming to clarify the feasibility and safety of use of low-dose dexmedetomidine for prevention of postoperative delirium in patients after intracranial operation for brain tumor.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients after elective intracranial operation for brain tumor under general anesthesia and who are admitted to the ICU directly from the operating room or postoperative care unit.

Exclusion Criteria:

* age under 18 years;
* admitted to the ICU after 22:00 PM;
* medical records documented preoperative history of mental or cognitive disorders including schizophrenia, epilepsy, Parkinsonism, or dementia;
* medical records documented inability to communicate in the preoperative period due to coma or language barrier;
* history of drug abuse of psychoactive and anesthetic drugs;
* known preoperative severe bradycardia (lower than 50 beats/min), sick sinus syndrome, second- or third-degree atrioventricular block, or left ventricular ejection fraction lower than 30%;
* serious hepatic dysfunction defined as Child-Pugh class C;
* severe renal dysfunction requiring renal replacement therapy before the surgery;
* allergies to ingredients or components of dexmedetomidine hydrochloride;
* American Society of Anesthesiologists classification of IV to VI;
* moribund condition with low likelihood of survival for more than 24 hours;
* pregnancy or lactation women;
* current enrollment in another clinical trial;
* refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Incidence of study agent interruption during the study | From the start of study agent infusion to postoperative day 1
  Predicted adverse events in the present study included bradycardia (defined as heart rate lower than 50 beats/min), hypotension (defined as systolic blood pressure lower than 90 mmHg), tachycardia (defined as heart rate greater than 100 beats/min), hypertension (defined as systolic blood pressure greater than 160 mmHg) and hypoxemia (defined as pulse oxygen saturation lower than 90%). The treatment of adverse events was determined by the responsible attending ICU physicians, who could stop the study agent infusion when the treatment failure or other conditions deemed necessary.

SECONDARY OUTCOMES:
Time from the end of operation to randomization | From the end of operation until the randomization, assessed up to 24 hours
  Time from the end of operation to randomization
Duration of study agent infusion | From the start of study agent infusion to postoperative day 1
  Duration of study agent infusion
Incidence of adverse events from the start of study agent infusion until 24 hours or until ICU discharge | From the start of study agent infusion to postoperative day 1
  Include bradycardia (defined as heart rate lower than 55 beats/min), hypotension (defined as systolic blood pressure lower than 90 mmHg), and hypoxemia (defined as pulse oxygen saturation lower than 90%)
Non-delirium complications | From the start of study agent infusion to postoperative day 28
  Include airway obstruction and apnea, respiratory failure, cardiac events, coma, epilepsy, cerebral hemorrhage or infarction, renal injury and infection

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Study Chair — Capital Medical University
Locations (1):
- ICU, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He X, Cheng KM, Duan YQ, Xu SS, Gao HR, Miao MY, Li HL, Chen K, Yang YL, Zhang L, Gu HQ, Zhou JX. Feasibility of low-dose dexmedetomidine for prevention of postoperative delirium after intracranial operations: a pilot randomized controlled trial. BMC Neurol. 2021 Dec 4;21(1):472. doi: 10.1186/s12883-021-02506-z. PMID 34863109